CLINICAL TRIAL: NCT01681797
Title: Fluorescence Angiography With Fluobeam™ Camera (Fluoptics Company): Planning and Monitoring of Perforator Flaps
Brief Title: Fluorescence Angiography: Planning and Monitoring of Perforator Flaps
Acronym: AFLU
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped due to lack of inclusion
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DCIC/11/13
Record Dates: First submitted 2012-08-31; First posted 2012-09-10 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Reconstructive Surgery
Keywords: fluorescent angiography; reconstructive surgery; perforator flap
MeSH Terms: interventions — Fluorescein Angiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- add-on fluorescence angiography (Experimental): The surgeon will prescribe the usual morphological assessment of the proposed flap:
  * CT angiography for an anterolateral thigh flap or an epigastric inferior flap
  * A Doppler ultrasonography for a fibula flap.
  In addition to the usual radiological technique used to locate the perforating arteries, the patient will have a fluorescence angiography prior to surgery, another just after the end of surgery and then one every six hours during the next 4 days.
  Interventions: Device: Fluorescence angiography (Fluobeam™ imaging system developed by Fluoptics company)

INTERVENTIONS:
Device: Fluorescence angiography (Fluobeam™ imaging system developed by Fluoptics company) — Fluorescence angiography after intravenous injection of Infracyanine® (indocyanine green)
  Other Names: The device used in this study is the Fluobeam™ imaging system developed by the company Fluoptics.; the technique requires the injection of a tracer Infracyanine® (SERB pharmaceutical company)

SUMMARY:
The purpose of this study is to determine whether fluorescence angiography is an effectiveness technique for the localization of vascular perforators and their area of perfusion and for the postoperative monitoring of flap perfusion.

DETAILED DESCRIPTION:
Reconstructive surgery is intended to replace amputated anatomical regions by autologous tissue taken from distant locations: flaps. The goal is to restitute ad integrum with minimal sequelae. Among the flaps available, perforator flaps have the advantage of being highly plastic, large and can be taken from accessory vessels the loss of wich does not compromise the vitality of the sampling site. However their more variable anatomy requires irradiating preoperative morphological assessment (CT angiography) or a doppler ultrasonography that is not always performed by the surgeon himself and does not distinguish between muscle perforator and skin perforator.

Fluorescence angiography is a superficial exploration technique of vascularization. After intravenous injection of a tracer (indocyanine green ICG), fluorescence angiography provides useful surface angiographic imaging in real-time. It can also help in monitoring intraoperative and postoperative quality of vascular anastomoses. Although fluorescence angiography has numerous applications (ophthalmology, neurosurgery, liver transplantation...), its usefulness in surgical flaps is only supported by a few publications. None really validate its clinical value by comparing it to reference investigations (CT angiography or doppler ultrasonography).

40 candidate for reconstructive surgery will be included in this study. The day before surgery, in addition to the usual technique used to locate perforator flaps, the patient will receive an injection of 0.025 mg / kg Infracyanine® (indocyanine green) and the area of interest of the flap will be explored with the Fluobeam™ camera.

Two hours after the surgery, during the usual clinical monitoring of the vitality of the flap, a new injection of Infracyanine® will test perfusion of the flap by measuring fluorescence intensity of the target area. These measurement will then be repeated every 6 hours for 4 days.

ELIGIBILITY:
Inclusion Criteria:

* perforator flap reconstruction whatever the indication (cancer, trauma, malformations). The main targets are the fibula flaps, anterolateral thigh flaps and inferior epigastric flaps
* consenting patient

Exclusion Criteria:

* known indocyanine green allergy
* pregnant woman, parturient woman or nursing woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-08; Primary Completion 2015-10-10 (Actual); Study Completion 2015-10-10 (Actual)

PRIMARY OUTCOMES:
Comparison between the position of perforator flap determined by fluorescence angiography and the real anatomic position of the flap determined after dissection | During the first fluorescent angiography
  For each flap, the position of the flap determined by fluorescent angiography will be compared with the anatomic position (actual) determined on the relevant flap after dissection (gold standard).

SECONDARY OUTCOMES:
Comparison between the position of the perforator flap determined by fluorescence angiography and the position of the flap determined by reference imaging techniques relevant to the flap (CT angiography or doppler ultrasonography) | During the first fluorescent angiography
  For each flap, the position of the flap determined by fluorescent angiography will be compared with the position determined by reference imaging techniques relevant to the flap (CT angiography or doppler ultrasonography)
Intraoperative monitoring of the quality of micro-vascular anastomoses using fluorescent angiography | Just after micro-vascular anastomoses
  Intraoperative monitoring of vascular flow through the micro-anastomoses will be determined by:
  * measuring the arterial and venous trans-anastomotic flow (ml / mm)
  * flow measurement (ml / mm) of an equivalent diameter vessel located in the operative field and not affected by the anastomosis
  * intrinsic transit time (in seconds) which is the time required for the fluorescence between the arterial anastomosis and the venous anastomosis
  * the number of leaks around the anastomosis.
Postoperative monitoring of flap perfusion using fluorescence angiography | Every six hours for four days after surgery
  This is to test the hypothesis that the dynamics of the fluorescence intensity in the area of interest is a prognostic factor for postoperative complications.

CONTACTS AND LOCATIONS:
Overall Officials: Georges BETTEGA, MD, PHD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital of Grenoble, Grenoble, Isere, France

REFERENCES:
- [Background] Koenig A, Herve L, Gonon G, Josserand V, Berger M, Dinten JM, Boutet J, Peltie P, Coll JL, Rizo P. Fluorescence diffuse optical tomography for free-space and multifluorophore studies. J Biomed Opt. 2010 Jan-Feb;15(1):016016. doi: 10.1117/1.3309738. PMID 20210462